CLINICAL TRIAL: NCT05935475
Title: A Comparative Study Between Electrocardiography Guided Technique Versus Anatomical Based Technique for Ideal Positioning of Dialysis Catheter Tip in Pediatric Patients
Brief Title: A Comparative Study for Ideal Positioning of Dialysis Catheter Tip in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sara Mabrouk Elghoul, Principal Investigator, Clinical lecturer of Pediatric Nephrology, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264PR196/5/23
Record Dates: First submitted 2023-06-20; First posted 2023-07-07 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Dialysis Catheter; Malposition

STUDY DESIGN:
Intervention Model Description: 150 children and adolescents with end stage renal disease or any cause for urgent hemodialysis at our nephrology Unit at TUH during the period of the study and classified into two equal groups: Group A (control): insertion of dialysis catheter using the anatomical landmark-guided technique.
  Group B: insertion of dialysis catheter using the ECG-guided technique.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be randomly assigned using an internet-based computer program (http://www.randomizer.org) either to the anatomical landmark group or to the ECG group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Active Comparator): 75 children and adolescent will insert dialysis catheter using the anatomical landmark technique
  Interventions: Procedure: Anatomical landmark guided dialysis catheter insertion
- group B (Active Comparator): 75 children and adolescent will insert dialysis catheter using the ECG guided technique
  Interventions: Procedure: ECG guided dialysis catheter insertion

INTERVENTIONS:
Procedure: Anatomical landmark guided dialysis catheter insertion — .: Before insertion, the catheter depth was calculated from the insertion point to the catheter tip point (midway the vertical line from the clavicular head of sternocleidomastoid to inter nipple line.
  Other Names: ultrasound guided dialysis catheter insertion using anatomical method
  Arms: group A
Procedure: ECG guided dialysis catheter insertion — after inserting the dialysis catheter into right IJV, the guidewire will be then withdrawn until the tip to be exactly positioned at the entry of the Superior Vena Cava in the right atrium. This will be ECG guided: the p wave appears as biphasic wave in the RA then the catheter will be withdrawn at 0.5 cm intervals until the P-wave returned to a normal configuration. (At that point, the catheter will be secured at the skin with suture and dressed with a transparent dressing
  Other Names: ultrasound guided dialysis catheter insertion using ECG technique
  Arms: group B

SUMMARY:
This prospective study will be conducted to compare between the efficacy of both ECG-guided technique and anatomical landmark technique to detect the ideal positioning of dialysis catheter tip and whether it will decrease the radiation exposure or no?

DETAILED DESCRIPTION:
This study will be conducted on 150 children and adolescents with end stage renal disease or any cause for urgent hemodialysis at our nephrology Unit at TUH during the period of the study and classified into two equal groups:

Group A (control): insertion of dialysis catheter using the anatomical landmark-guided technique.

Group B: insertion of dialysis catheter using the ECG-guided technique. Participants will be randomly assigned using an internet-based computer program (http://www.randomizer.org) either to the anatomical landmark group or to the ECG group.

All patients included in the study will be subjected to:

1. History taking including the cause of dialysis.
2. Clinical examination.
3. Investigations:

   * Complete blood picture
   * Bleeding and clotting time.
   * International normalized ratio
   * Serum potassium
   * Serum creatinine, blood urea level.
4. Procedure technique:

A single anesthiologist will perform the procedures in both groups under complete a septic condition after consent taking from the child guardians. All participants will be cannulated in the right internal jugular vein (IJV). The participants were placed in Trendelenburg position and the dialysis catheter will be inserted using catheter-over-guidewire technique (the Seldinger technique) with the aid of ultrasound for scanning the neck by the superficial probe (7-13 MHz).

In the ECG-guided technique, after inserting the dialysis catheter into right IJV, the guidewire will be then withdrawn until the tip to be exactly positioned at the entry of the Superior Vena Cava in the right atrium. This will be ECG guided: the p wave appears as biphasic wave in the RA then the catheter will be withdrawn at 0.5 cm intervals until the P-wave returned to a normal configuration. At that point, the catheter will be secured at the skin with suture and dressed with a transparent dressing.

In the anatomical landmark technique: Before insertion, the catheter depth was calculated from the insertion point to the catheter tip point (midway the vertical line from the clavicular head of sternocleidomastoid to inter nipple line.

After insertion of the dialysis catheter, the patient will be monitored for any hemodynamic deterioration and a repeat ultrasound-chest was done to rule out pneumothorax. An anterior-posterior CXR in supine position will be taken in all patients, to confirm the placement and positioning of the dialysis catheter.

The whole length of the SVC was defined on CXR as the area from the lower border on the first right costal cartilage close to the sternum to the conventional radiographic SVC-RA junction.

Post insertion CXR done in both groups to detect the adequate insertion length of the dialysis catheter, frequency of CXR for repositioning, time to dialysis catheter placement, and post procedural complications will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients from 5 to 18 years require dialysis catheter insertion for any indication as acute or chronic renal failure.

Exclusion Criteria:

* Patients with coagulopathy.
* Patients with infection.
* Patients with cardiac arrhythmia or pacemaker

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2023-05-28 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
The ideal tip position of dialysis catheter | one year
  all the participant will be cannulated in the right internal jugular vein by the Seldinger technique with the aid of ultrasound, In the ECG-guided technique,the wire will be withdrawn until positioned at the entry of the Superior Vena Cava in the right atrium and the P-wave returned to a normal configuration.In the anatomical landmark technique: Before insertion, the catheter depth was calculated from the insertion point to a point (midway the vertical line from the clavicular head of sternocleidomastoid to inter nipple line.An anterior-posterior CXR in supine position will be taken in all patients, to confirm the placement and positioning of the dialysis catheterThe whole length of the SVC was defined on CXR as the area from the lower border on the first right costal cartilage close to the sternum to the conventional radiographic SVC-RA junction

SECONDARY OUTCOMES:
Post insertion adverse events | one year
  After insertion of the dialysis catheter, the patient will be monitored for any hemodynamic deterioration and a repeat ultrasound-chest was done to rule out pneumothorax.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Mabrouk Mohamed Elghoul, Principal Investigator — Tanta University
Locations (1):
- Sara Mabrouk Mohamed Elghoul, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No
no individual participant data will be shared